CLINICAL TRIAL: NCT02782598
Title: The Application of Negative Atrioventricular Hysteresis in Cardiac Resynchronization Therapy With MultiPoint Pacing
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD_856
Record Dates: First submitted 2016-05-19; First posted 2016-05-25 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
Keywords: Negative; Atrioventricular; Hysteresis; Cardiac Resynchronization; MultiPoint
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRT+NAVH: Surface ECG and pressure-volume loop recordings will be taken during the adjustment of programmable Cardiac Resynchronization Therapy and Negative Atrioventricular Hysteresis settings at the device implant procedure
  Interventions: Device: CRT+NAVH

INTERVENTIONS:
Device: CRT+NAVH — Cardiac Resynchronization Therapy with Negative Atrioventricular Hysteresis

SUMMARY:
The purpose of this study is to evaluate the application of Negative AV Hysteresis (NAVH) to improve electrical synchrony in MultiPoint Pacing (MPP) Cardiac Resynchronization Therapy (CRT) patients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for implantation of an MPP-enabled SJM Quadripolar CRT Pacing System
* QRS duration > 140 ms
* Left bundle branch block documented
* Ability to provide informed consent for study participation
* Willing to comply with the study evaluation requirements
* At least 18 years of age

Exclusion Criteria:

* Resting ventricular rate >100 bpm
* Intrinsic PR interval > 300 ms
* Paroxysmal or persistent atrial tachycardia or atrial fibrillation documented
* A recent myocardial infarction, ablation, drug intoxication, electrolyte imbalance, or any condition within the last 90 days that would be contraindicated for CRT programming changes in the opinion of the investigator
* Women who are pregnant or who plan to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment will include patients scheduled to be implanted with MultiPoint Pacing-enabled SJM Quadripolar Pacing Systems
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Acute change in QRS duration due to CRT with NAVH, relative to intrinsic conduction | 1 day
  Acute changes in surface ECG QRS duration resulting from Cardiac Resynchronization Therapy (CRT) with Negative Atrioventricular Hysteresis (NAVH) over a range of programmable values

SECONDARY OUTCOMES:
Acute changes in LV pressure-volume hemodynamics due to CRT with NAVH, relative to intrinsic conduction | 1 day
  Acute changes in left ventricular pressure-volume hemodynamics resulting from Cardiac Resynchronization Therapy with Negative Atrioventricular Hysteresis over a range of programmable values
Change in QRS duration after one day of CRT with NAVH, relative to intrinsic conduction | 1 day
  Changes in surface ECG QRS duration after one day of Cardiac Resynchronization Therapy with Negative Atrioventricular Hysteresis

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, MI, Italy